CLINICAL TRIAL: NCT07016698
Title: A Prospective, Multicenter, Single Arm, Real-World Registry Assessing the Clinical Use of the Rotarex(TM) Rotational Excisional Atherectomy System (XTRACT Registry)
Brief Title: Real-World Registry of the Rotarex(TM) Rotational Excisional Atherectomy System (XTRACT Registry)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDPI-25-001
Record Dates: First submitted 2025-05-28; First posted 2025-06-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Arterial Disease(PAD)
Keywords: Rotarex; PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Rotarex(TM) Rotational Excisional Atherectomy System (Other): Subjects treated with RotarexTM Rotational Excisional Atherectomy System
  Interventions: Device: Rotarex(TM) Rotational Excisional Atherectomy System

INTERVENTIONS:
Device: Rotarex(TM) Rotational Excisional Atherectomy System — Subjects treated with Rotarex(TM) Rotational Excisional Atherectomy System

SUMMARY:
The XTRACT Registry is a prospective, single arm multicenter study on the use of on the Rotarex(TM) Rotational Excisional Atherectomy System.

DETAILED DESCRIPTION:
The study will recruit approximately 600 subjects treated for PAD.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legally authorized representative provides written informed consent using an Informed Consent Form (ICF) that is reviewed and approved by the IRB for the site.
2. Subject is ≥22 years old at the time of signing the informed consent.
3. Subject must have a lesion(s) in their infra-inguinal peripheral arteries that can be treated with the RotarexTM Rotational Excisional Atherectomy System according to Instructions For Use (IFU).
4. Rutherford 2-5 for chronic limb ischemia and Rutherford I to IIb for acute limb ischemia.
5. Target lesion can be crossed intra-luminally by guidewire.
6. At least one patent native outflow artery to the foot, free from significant stenosis(≥50% stenosis as confirmed by angiography) (ChLI Cohort only, not applicable to ALI Cohort).

Exclusion Criteria:

1. Subject is unable or unwilling to comply with follow-up procedures and visits.
2. Subject has a target lesion in a vessel with less than 3 mm in diameter.
3. Subject is participating in another device or drug clinical trial that interferes with this protocol and confounds results.
4. Treatment plan includes use of a thrombectomy and/or atherectomy device other than RotarexTM Rotational Excisional Atherectomy System.
5. Life expectancy is below 1 year.
6. Pregnant, planning to become pregnant during the course of the study or nursing a child.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | Immediate Post Index Procedure
  Procedural Success defined as the rate of successful revascularization of target lesion (residual stenosis/thrombus ≤30%) following index procedure.
Freedom from major complications | 30 days post index procedure
  Freedom from composite of device and/or procedure related perioperative (≤30 day) death, unplanned target limb major amputation (above the ankle), and clinically driven target lesion revascularization (CD-TLR) at 30 days post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Krishnan, MD, FACC, Principal Investigator — The Icahn School of Medicine, The Mount Sinai Health System; Todd L Berland, MD, FACS, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Radiology and Imaging Specialists, Lakeland, Florida
  - Vital Heart and Vein, Humble, Texas

IPD SHARING:
Plan to Share IPD: No